CLINICAL TRIAL: NCT03532581
Title: A Novel Surgical Technique: Indocyanine Green Lymphangiography for Identification of the Thoracic Duct During Neck Dissection
Brief Title: Indocyanine Green Lymphangiography in Identifying Thoracic Duct During Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, John Phay, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-17368; NCI-2018-00390 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-04-19; First posted 2018-05-22 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Neck Dissection; Radical Lymph Node Dissection
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (ICG lymphangiography) (Experimental): Participants receive indocyanine green solution SC and undergo near-infrared imaging over 1-2 minutes during their standard of care neck surgery.
  Interventions: Other: Indocyanine Green Solution; Procedure: Lymphangiography

INTERVENTIONS:
Other: Indocyanine Green Solution — Given Subcutaneous injection
  Other Names: IC-GREEN; ICG Solution
Procedure: Lymphangiography — Undergo lymphangiography
  Other Names: Lymphography

SUMMARY:
This phase I trial studies how well indocyanine green lymphangiography works in identifying thoracic duct during neck surgery. Diagnostic procedures, such as near infrared fluorescence imaging with indocyanine green may help recognize and prevent injury to thoracic duct during neck surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Feasibility and optimization of thoracic duct identification using indocyanine green (ICG) lymphangiography.

II. To explore specifically how identifying the thoracic duct (TD) will prevent injury intra-operatively.

III. To understand if a TD injury can be recognized by leakage of fluorescent chyle into the operating field.

OUTLINE:

Participants receive indocyanine green solution subcutaneously (SC) and undergo near-infrared imaging over 1-2 minutes during their standard of care neck surgery.

After completion of study treatment, participants are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients who are undergoing LEFT modified radical or selective (including zone IV) lymph node dissection for any indication; this includes patients who have had prior neck surgery

Exclusion Criteria:

* Children, minors, pregnant women, women who are breast feeding, institutionalized patients
* Known prior allergic reaction to ICG or allergy to iodine
* Patients with excessively high anesthesia risks who cannot tolerate the extra time under general anesthesia needed to perform this study; the surgeon and anesthesiologist will determine this pre-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Identify thoracic duct (TD) using indocyanine green (ICG) | Up to 1 year
  We will determine in how many patients the thoracic duct is identified by white light visualization and by ICG fluorescence. The collected data will be primarily qualitative as determined by the surgeon.
Prevent injury to the TD | Up to 1 year
  Percentage of patients with TD injury will be calculated and compared to contemporary rates of injury.
Recognize injury intra-operatively | Up to 1 year
  Will be mostly qualitative data collection on how the injury was identified and in what percent.

CONTACTS AND LOCATIONS:
Overall Officials: John Phay, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu